CLINICAL TRIAL: NCT01473836
Title: A Phase 3, Multicenter, Unblind, Non-Comparative Study To Confirm Efficacy And Safety Of Intravenous Metronidazole In Patients With Intrabdominal Infection In Combination With Intravenous Ceftriaxone
Brief Title: A Phase 3 Study Of Intravenous Metronidazole For Intrabdominal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6831005
Record Dates: First submitted 2011-10-11; First posted 2011-11-17 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Intra-abdominal Infections
Keywords: Metronidazole; intra-abdominal infection; pelvic inflammatory disease; anaerobe
MeSH Terms: conditions — Intraabdominal Infections; Pelvic Inflammatory Disease | interventions — Metronidazole; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metronidazole (Experimental): Metronidazole will be administered at a dose of 500 mg TID (or QID for refractory or severe infection) in combination with ceftriaxone sodium
  Interventions: Drug: Metronidazole; Drug: Ceftriaxone sodium

INTERVENTIONS:
Drug: Metronidazole — Metronidazole will be administered at a dose of 500 mg TID (or QID for refractory or severe infection) for 3 to 14 days, in principle. Treatment duration can be prolonged up to 21 days based on subject's condition.
Drug: Ceftriaxone sodium — Ceftriaxone sodium will be administered at a daily dose of 2 g (strength) when metronidazole is administered TID or at a daily dose of 4 g (strength) when metronidazole is administered QID.
  Other Names: ROCEPHIN

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety in Japanese adult subjects with Intra-abdominal/Pelvic infections receiving Metronidazole IV 1,500-2,000 mg/day in combination with ceftriaxone sodium.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older.
* Diagnosed with intra-abdominal infections or pelvic inflammatory diseases.
* Can be obtained a specimen for bacteriological efficacy assessment.

Exclusion Criteria:

* Known or suspected hypersensitivity, intolerance or contraindication to Metronidazole, Ceftriaxone sodium, or other cephem antibiotics.
* Severe renal dysfunction (creatinine clearance < 30 mL/min.) Reference: Cockcroft-Gault calculation formula.
* Hepatic dysfunction (AST, ALT, total bilirubin > 3 times upper limit of normal range values).
* Severe underlying disease; patients in which drug clinical evaluation is difficult because of confounding diseases.

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Japan (15):
  - Daiyukai First Hospital, Ichinomiya, Aichi-ken
  - Hirosaki National Hospital, Hirosaki, Aomori
  - National Hospital Organization Chiba Medical Center, Chiba, Chiba
  - National Hospital Organization Kokura Medical Center, Kitakyushu, Fukuoka
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Kawasaki Saiwai Hospital, Kawasaki, Kanagawa
  - Kumamoto Saishunso National Hospital, Koushi, Kumamoto
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Iida Municipal Hospital, Iida, Nagano
  - Nagano Prefectural Suzaka Hospital, Suzaka-shi, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ohmura, Nagasaki
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Koshigaya Municipal Hospital, Koshigaya, Saitama

REFERENCES:
- [Derived] Mikamo H, Matsumizu M, Nakazuru Y, Nagashima M. Efficacy and safety of metronidazole injection for the treatment of infectious peritonitis, abdominal abscess and pelvic inflammatory diseases in Japan. J Infect Chemother. 2015 Feb;21(2):96-104. doi: 10.1016/j.jiac.2014.10.005. Epub 2014 Nov 28. PMID 25442806
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6831005&StudyName=A%20Phase%203%20Study%20Of%20Intravenous%20Metronidazole%20For%20Intrabdominal%20Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- Metronidazole/Ceftriaxone: Metronidazole was administered in combination with ceftriaxone sodium, at a dose of 500 mg three times a day (TID) or four times a day (QID) for refractory or severe infection. Ceftriaxone was administered at the dose of 1 g twice a day (BID) when metronidazole was administered TID, or at dose of 2 g BID when metronidazole was administered QID. The duration of drug administration was 3 to 14 days.
Period: Overall Study
Arm/Group | Metronidazole/Ceftriaxone
Started | 38
Completed | 32
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Does not meet entrance criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response: Response Rate (Data Review Committee Assessment)
Description: Clinical response was evaluated by the data review committee as effective (cured or improved), ineffective (not meeting "effective" criteria), or indeterminate at the end of treatment (EOT) and the test of cure (TOC: 7 days after EOT) based on clinical symptoms, ultrasound images and necessity of other treatment. TOC was the primary analysis of this outcome measure. Cured = clinical symptoms and abnormal findings at the start of the study were disappeared and considered other antibiotics were not required during the study and after the assessment time point. Improved = clinical symptoms and abnormal findings at the start of the study were improved and considered other antibiotics were not required during the study and after the assessment time point. Response rate was calculated from the following formula; "number of participants evaluated as effective" over "total number of participants that excluding ones evaluated as indeterminate" multiplied by 100.
Time Frame: Baseline to EOT (up to 14 days), TOC
Population: Clinical per protocol set consisted of all participants who received at least one dose of study medication, had no significant protocol deviation, and underwent planned assessments. No imputation was used for missing data. n = number of participants assessed that excluding ones evaluated as "indeterminate".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 30
percentage of participants
  End of Treatment (n=30) | 96.6 [82.2 to 99.9]
  Test of Cure (n=30) | 96.7 [82.8 to 99.9]

2. Secondary Outcome: Clinical Response: Response Rate (Investigator Assessment)
Description: Clinical response was evaluated by the investigator as effective (cured or improved), ineffective (not meeting "effective" criteria), or indeterminate at the end of treatment (EOT) and the test of cure (TOC: 7 days after EOT) based on clinical symptoms, ultrasound images and necessity of other treatment. TOC was the primary analysis of this outcome measure. Cured = clinical symptoms and abnormal findings at the start of the study were disappeared and considered other antibiotics were not required during the study and after the assessment time point. Improved = clinical symptoms and abnormal findings at the start of the study were improved and considered other antibiotics were not required during the study and after the assessment time point. Response rate was calculated from the following formula; "number of participants evaluated as effective" over "total number of participants that excluding ones evaluated as indeterminate" multiplied by 100.
Time Frame: Baseline to EOT (up to 14 days), TOC
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 30
percentage of participants
  End of Treatment (n=30) | 96.7 [82.8 to 99.9]
  Test of Cure (n=29) | 100.0 [88.1 to 100.0]

3. Secondary Outcome: Percentage of Participants Who Was Assessed as Appropriate to Continue Treatment (Investigator Assessment)
Description: The appropriateness of treatment continuation was evaluated on Day 4 by the investigator as continuation, discontinuation or indeterminate based on the clinical response. The percentage of participants was calculated from the following formula; "number of participants assessed as continuation" over "total number of participants that excluding ones assessed as indeterminate" multiplied by 100.
Time Frame: Baseline to Day 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 30
percentage of participants | 100.0

4. Secondary Outcome: Bacteriological Response: Eradication Rate (Data Review Committee Assessment)
Description: Bacteriological response was evaluated as eradication (eradication, presumed eradication or colonization), persistence, or indeterminate by the data review committee, at Day 4, at the end of treatment (EOT), and the test of cure (TOC: 7 days after EOT). Eradication Rate was calculated from the following formula, "number of participants with bacteria eradication, presumed eradication or colonization" over "total number of participants that excluding ones evaluated as indeterminate" multiplied by 100.
Time Frame: Baseline to Day 4, EOT (up to 14 days), TOC
Population: Bacteriologic per protocol set consisted of all participants in the clinical per protocol set in whom bacterial pathogens were identified on Day 1 prior to the initial dose. No imputation was used for missing data. n = number of participants assessed that excluding ones evaluated as "indeterminate".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 21
percentage of participants
  Day 4 | 100.0 [75.3 to 100.0]
  End of Treatment | 100.0 [83.2 to 100.0]
  Test of Cure | 100.0 [83.9 to 100.0]

5. Secondary Outcome: Bacteriological Response: Eradication Rate (Investigator Assessment)
Description: Bacteriological response was evaluated as eradication (eradication, presumed eradication or colonization), persistence, or indeterminate by the investigator at the end of treatment (EOT), and the test of cure (TOC: 7 days after EOT). Eradication Rate was calculated from the following formula, "number of participants with bacteria eradication, presumed eradication or colonization" over "total number of participants that excluding ones evaluated as indeterminate" multiplied by 100.
Time Frame: Baseline to Day 4, EOT (up to 14 days), TOC
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 21
percentage of participants
  Day 4 | 100.0 [75.3 to 100.0]
  EOT | 100.0 [83.2 to 100.0]
  TOC | 100.0 [83.9 to 100.0]

6. Secondary Outcome: Number of Participants Analyzed for Population Pharmacokinetics (PK) of Metronidazole
Description: Population pharmacokinetic analysis of Metronidazole is conducted by combining current study data with other Metronidazole studies.
Time Frame: Four samples were taken at any infusion after the first dosing: during infusion, immediately after end of infusion, between 15 and 60 minutes after end of infusion, and between 2 hours and immediately before the start of the next infusion.
Population: No population pharmacokinetic analysis results are available just for the current study.
Arm/Group | Metronidazole/Ceftriaxone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Metronidazole/Ceftriaxone
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 30/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metronidazole/Ceftriaxone (N=38)
Infectious peritonitis (Infections and infestations) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metronidazole/Ceftriaxone (N=38)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 12
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Injection site extravasation (General disorders) | 1
Injection site pain (General disorders) | 3
Instillation site erythema (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Injection site infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood potassium increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Dysuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.